CLINICAL TRIAL: NCT00060723
Title: Behavioral Effect of Obstructive Sleep Apnea in Children
Brief Title: Behavioral Effects of Obstructive Sleep Apnea in Children
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ronald D. Chervin, M.D., M.S., Michael S Aldrich Collegiate Professor of Sleep Medicine and Professor of Neurology, University of Michigan
Other Study IDs: 5R01HD38461-3; 5R01HD038461 (NIH)
Record Dates: First submitted 2003-05-09; First posted 2003-05-13 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Sleep-disordered Breathing; Sleep Apnea, Obstructive; ADHD
Keywords: Polysomnography; Sleep-disordered breathing; Sleep apnea, obstructive; Hyperactivity; Sleep; Child
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adenotonsillectomy group: Children ages 5-12 who are scheduled for adenotonsillectomy for obstructive sleep apnea
- Comparison group: Children ages 5-12, scheduled for hernia repairs, other procedures not involving the head, chest or neck, or no procedures. Additional exclusions include children with a history of recurrent throat infections, large tonsils, history of or plans for adenoidectomy and/or tonsillectomy or who have been previously diagnosed with sleep-disordered breathing.

SUMMARY:
Sleep-disordered breathing (SDB) in children may be responsible for disruptive daytime behaviors such as inattention and hyperactivity. Many children undergo tonsillectomy for SDB and disruptive daytime behaviors. However, the link between SDB and disruptive behavior is not clearly understood. This study will evaluate the relationship between SDB and disruptive behavior.

DETAILED DESCRIPTION:
While adenotonsillectomy (AT) remains one of the most common surgical procedures performed in children, indications for AT have changed in recent years. Surgeons now perform AT for suspected obstructive SDB and for daytime behaviors that may be a consequence of SDB, such as inattention and hyperactivity. However, whether SDB causes these and other disruptive behaviors is not well known. Further, the precise nature of these behaviors and what types or levels of SDB may be of concern are poorly understood. Consequently, pediatricians and otolaryngologists are not able to use objective preoperative testing to assess SDB and abnormal behavior.

This research project seeks to better define the relationship between childhood SDB and daytime behavioral problems and to determine whether SDB actually causes these behaviors. The study will better define whether inattention and hyperactivity are frequent among children who undergo AT, will identify measures and levels of SDB that are indicative of these behaviors, and will test whether improvement in SDB after AT is associated with improvement in behavior.

Five- to twelve-year-old children who have been scheduled for AT or for a control group procedure (minimally invasive, non-airway-related surgeries such as herniorraphies) will undergo behavioral assessments, cognitive tests, and structured psychiatric interviews. A secondary control group will include healthy children who are not scheduled for any type of surgery. Preoperative assessments will be used to define what behaviors are more prominent in the children scheduled for AT than in children scheduled for hernia repair. All children will undergo preoperative polysomnography to detect subtle forms of SDB that may be particularly prevalent in children. Children will also undergo assessments after surgery.

Children will be scheduled for two or three study visits, depending on whether participants agreed to an optional 3-month interim assessment. Children will be followed for approximately 1 year from the date of surgery.

ELIGIBILITY:
Inclusion Criteria

* Scheduled for adenotonsillectomy at participating local otolaryngology practices

Exclusion Criteria

* Serious health conditions that make interpretation of sleep studies or cognitive testing difficult
* Mental or physical handicaps that prevent proper interpretation of behavioral tests
* Current treatment by a physician for SDB
* Previous surgeries for SDB, such as adenoidectomy and/or tonsillectomy or other airway-related surgeries
* Inability to schedule sleep and behavioral testing prior to surgery
* Requires sleep or behavioral testing for clinical indications
* Planning to schedule additional surgeries within 1 year of study entry
* Unreliable or inconvenient access to the University of Michigan facilities within 1 year of study entry

Additional Exclusion Criteria for Control Group

* History of large, uninfected tonsils
* History of recurrent throat infections ( > 7 infections in one year, > 5 infections in each of two years, or > 3 infections in each of 3 years)
* History of adenoidectomy, tonsillectomy, or other treatment for SDB
* Planned adenoidectomy and/or tonsillectomy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric Otolaryngology surgery practices and primary care or general surgery practices at University of Michigan and St. Joseph Mercy Health Systems
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 1999-08; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Chervin, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- Univerisity of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Weatherly RA, Mai EF, Ruzicka DL, Chervin RD. Identification and evaluation of obstructive sleep apnea prior to adenotonsillectomy in children: a survey of practice patterns. Sleep Med. 2003 Jul;4(4):297-307. doi: 10.1016/s1389-9457(03)00100-x. PMID 14592302
- [Background] Chervin RD, Ruzicka DL, Wiebelhaus JL, Hegeman GL 3rd, Marriott DJ, Marcus CL, Giordani BJ, Weatherly RA, Dillon JE. Tolerance of esophageal pressure monitoring during polysomnography in children. Sleep. 2003 Dec 15;26(8):1022-6. doi: 10.1093/sleep/26.8.1022. PMID 14746385
- [Background] Archbold KH, Giordani B, Ruzicka DL, Chervin RD. Cognitive executive dysfunction in children with mild sleep-disordered breathing. Biol Res Nurs. 2004 Jan;5(3):168-76. doi: 10.1177/1099800403260261. PMID 14737917
- [Background] Chervin RD, Burns JW, Subotic NS, Roussi C, Thelen B, Ruzicka DL. Method for detection of respiratory cycle-related EEG changes in sleep-disordered breathing. Sleep. 2004 Feb 1;27(1):110-5. doi: 10.1093/sleep/27.1.110. PMID 14998246
- [Background] Chervin RD, Burns JW, Subotic NS, Roussi C, Thelen B, Ruzicka DL. Correlates of respiratory cycle-related EEG changes in children with sleep-disordered breathing. Sleep. 2004 Feb 1;27(1):116-21. doi: 10.1093/sleep/27.1.116. PMID 14998247
- [Result] Giordani B, Hodges EK, Guire KE, Ruzicka DL, Dillon JE, Weatherly RA, Garetz SL, Chervin RD. Changes in neuropsychological and behavioral functioning in children with and without obstructive sleep apnea following Tonsillectomy. J Int Neuropsychol Soc. 2012 Mar;18(2):212-22. doi: 10.1017/S1355617711001743. Epub 2012 Jan 25. PMID 22272653
- [Result] Giordani B, Hodges EK, Guire KE, Ruzicka DL, Dillon JE, Weatherly RA, Garetz SL, Chervin RD. Neuropsychological and behavioral functioning in children with and without obstructive sleep apnea referred for tonsillectomy. J Int Neuropsychol Soc. 2008 Jul;14(4):571-81. doi: 10.1017/S1355617708080776. PMID 18577286
- [Result] Dillon JE, Blunden S, Ruzicka DL, Guire KE, Champine D, Weatherly RA, Hodges EK, Giordani BJ, Chervin RD. DSM-IV diagnoses and obstructive sleep apnea in children before and 1 year after adenotonsillectomy. J Am Acad Child Adolesc Psychiatry. 2007 Nov;46(11):1425-36. doi: 10.1097/chi.0b013e31814b8eb2. PMID 18049292
- [Result] Chervin RD, Weatherly RA, Garetz SL, Ruzicka DL, Giordani BJ, Hodges EK, Dillon JE, Guire KE. Pediatric sleep questionnaire: prediction of sleep apnea and outcomes. Arch Otolaryngol Head Neck Surg. 2007 Mar;133(3):216-22. doi: 10.1001/archotol.133.3.216. PMID 17372077
- [Result] Chervin RD, Weatherly RA, Ruzicka DL, Burns JW, Giordani BJ, Dillon JE, Marcus CL, Garetz SL, Hoban TF, Guire KE. Subjective sleepiness and polysomnographic correlates in children scheduled for adenotonsillectomy vs other surgical care. Sleep. 2006 Apr;29(4):495-503. PMID 16676783
- [Result] Chervin RD, Ruzicka DL, Giordani BJ, Weatherly RA, Dillon JE, Hodges EK, Marcus CL, Guire KE. Sleep-disordered breathing, behavior, and cognition in children before and after adenotonsillectomy. Pediatrics. 2006 Apr;117(4):e769-78. doi: 10.1542/peds.2005-1837. PMID 16585288